CLINICAL TRIAL: NCT05839405
Title: Food Allergy in the Brain: Investigating the Impact of Food Allergy on Children's Mental Health and Cognition, and the Associated Neurobiological Mechanisms
Brief Title: Food Allergy in the Brain
Acronym: FAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 322589
Record Dates: First submitted 2023-02-27; First posted 2023-05-03 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-02

CONDITIONS: Food Allergy; Food Allergy in Children; Anxiety; Cognitive Symptom
MeSH Terms: conditions — Food Hypersensitivity; Anxiety Disorders; Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non Allergic: Recruited patients whose medical records indicate they are not allergic to the foods they were in clinic for
  Interventions: Other: None - Cross Sectional.
- Mild Allergic: Recruited patients whose medical records indicate they are allergic to the foods they were in clinic for, but only to a mild degree where they would be expected to experience mild, non-life threatening symptoms on exposure to the allergen
  Interventions: Other: None - Cross Sectional.
- Severe Allergic: Recruited patients whose medical records indicate they are allergic to the foods they were in clinic for, to a severe degree where they would be expected to experience severe symptoms on exposure to the allergen
  Interventions: Other: None - Cross Sectional.

INTERVENTIONS:
Other: None - Cross Sectional. — There is no intervention, this is cross-sectional only.

SUMMARY:
Preventing food allergic reactions predominantly relies on allergen avoidance and managing this daily causes high anxiety in some patients, while having an allergic reaction can cause a post-traumatic stress disorder-like syndrome in children. The underlying mechanisms of these psychological changes are poorly understood, but one potential mechanism may be post-natal hippocampal neurogenesis (HN). HN is the production of new neurons from stem cells in the hippocampus which is one of the brain centres for memory and mood regulation. HN has been associated with cognitive function and some psychiatric disorders. Importantly, it can be influenced by both internal (bloodstream) and external (exercise, diet, etc.) factors. This study will explore the link between food allergy and children's mental health and cognition, and to determine whether this is linked to changes in HN.

DETAILED DESCRIPTION:
Preventing food allergic reactions predominantly relies on allergen avoidance and managing this daily causes high anxiety in some patients, while having an allergic reaction can cause a post-traumatic stress disorder-like syndrome in children. The underlying mechanisms of these psychological changes are poorly understood, but one potential mechanism may be post-natal hippocampal neurogenesis (HN). HN is the production of new neurons from stem cells in the hippocampus which is one of the brain centres for memory and mood regulation. HN has been associated with cognitive function and some psychiatric disorders. Importantly, it can be influenced by both internal (bloodstream) and external (exercise, diet, etc.) factors. This study will explore the link between food allergy and children's mental health and cognition, and to determine whether this is linked to changes in HN.

This study will recruit child patients (aged 8-15 years), and their legal parent/guardian, that are attending a routine clinic appointment at the Paediatric Allergy Unit at St Thomas' Hospital. Parent/guardians and the child will be approached by the patient's direct clinical team, who will explain the study procedures involved in participation. Consented adult (parent/guardian) participants will be asked to complete three anxiety questionnaires, to assess the influence of parental anxiety on that of the child. Consented child participants will be asked to complete two anxiety questionnaires and a memory task. Blood samples from the patient will also be collected in addition to those taken as part of their routine clinic appointment. Specifically, blood will be collected in the following tubes: gold top Vacutainer tube containing clot activator and gel for serum separation (4ml 8-15yrs), green top Vacutainer tube containing lithium heparin for whole blood (4ml 8-15yrs), and blue top Vacutainer tube containing citrate for peripheral blood mononuclear cell (PBMC) and plasma separation and storage (30ml 8-12yrs; 50ml 13-15yrs).

The plasma and serum from this collection will be used on two stem cell models that mimic food allergic reactions and HN, respectively. Any differences in these processes will be analysed alongside the questionnaire and memory task data and, if a link is successfully demonstrated, further work will aim to identify blood-borne factors responsible for these changes. This study will shed light on the impact of food allergy on children's mental health as well as the biological processes behind it.

ELIGIBILITY:
Inclusion Criteria:

* • Children ≥ 8 years old and <16 years

  * Suspected food allergy (non-defined allergen)
  * Undergoing blood collection for IgE testing at their clinic appointment
  * Fluent / age-appropriate level of English (verbal and written) of both the child and legal parent / guardian

Exclusion Criteria:

* Diagnosed neurological disorders and learning disabilities, including autism spectrum disorder, attention deficit hyperactivity disorder, Down's Syndrome.

  * Undergoing any allergen-specific immunotherapy or other immunomodulatory treatments such as biologics and immunosuppressants

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will recruit child patients (aged 8-15 years), and their legal parent/guardian, that are attending a routine clinic appointment at the Paediatric Allergy Unit at St Thomas' Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of DAPI-positive cells by allergic group | Throughout study, on average 2.5 years
  After exposure to patient serum, the number of DAPI-positive cells will be measured in the in vitro assay will be measured
%Ki67-positive cells by allergic group | Throughout study, on average 2.5 years
  After exposure to patient serum, cells fluorescently expressing Ki67 will be quantified within a total pool of cells that are fluorescently positive for DAPI (a nuclear DNA stain), i.e., total percentage of double fluorescently labelled cells within a total single (DAPI) stained population.
%CC3-positive cells by allergic group | Throughout study, on average 2.5 years
  After exposure to patient serum, cells fluorescently expressing CC3 will be quantified within a total pool of cells that are fluorescently positive for DAPI (a nuclear DNA stain), i.e., total percentage of double fluorescently labelled cells within a total single (DAPI) stained population.
%Nestin-positive cells by allergic group | Throughout study, on average 2.5 years
  After exposure to patient serum, cells fluorescently expressing Nestin will be quantified within a total pool of cells that are fluorescently positive for DAPI (a nuclear DNA stain), i.e., total percentage of double fluorescently labelled cells within a total single (DAPI) stained population.
%SOX2-positive cells by allergic group | Throughout study, on average 2.5 years
  After exposure to patient serum, cells fluorescently expressing SOX2 will be quantified within a total pool of cells that are fluorescently positive for DAPI (a nuclear DNA stain), i.e., total percentage of double fluorescently labelled cells within a total single (DAPI) stained population.
%MAP2-positive cells by allergic group | Throughout study, on average 2.5 years
  After exposure to patient serum, cells fluorescently expressing MAP2 will be quantified within a total pool of cells that are fluorescently positive for DAPI (a nuclear DNA stain), i.e., total percentage of double fluorescently labelled cells within a total single (DAPI) stained population.
%DCX-positive cells by allergic group | Throughout study, on average 2.5 years
  After exposure to patient serum, cells fluorescently expressing DCX will be quantified within a total pool of cells that are fluorescently positive for DAPI (a nuclear DNA stain), i.e., total percentage of double fluorescently labelled cells within a total single (DAPI) stained population.

SECONDARY OUTCOMES:
General anxiety levels of children by their allergic status, using the Spence's Children's Anxiety Scale | Throughout study, on average 2.5 years
  To determine whether food allergy is associated with changes to general anxiety in children. General anxiety levels will be assessed using the Spence's Children's Anxiety Scale, which has a minimum value of 0 and a maximum value of 114, with higher scores indicating higher levels of anxiety. Mean anxiety scores will be compared across allergic groups.
General anxiety levels of parents by their child's allergic status, using the Hospital Anxiety Depression Scale | Throughout study, on average 2.5 years
  To determine whether food allergy is associated with changes to general anxiety in the legal caregiver. General anxiety levels will be assessed using the Hospital Anxiety Depression Scale, which has a minimum limit of 0 and a maximum limit of 21 for anxiety, with a higher score representing higher levels of anxiety. Mean anxiety scores will be compared across allergic groups. Mean anxiety scores will be compared across allergic groups.
Food allergy-specific anxiety levels of children by their allergic status, using the Worry About Food Allergy scale | Throughout study, on average 2.5 years
  To determine whether food allergy is associated with changes to food allergy-specific anxiety in children. Food allergy-specific anxiety levels in children will be assessed using the Worry About Food Allergy Child (8-12yrs) and Teen scales (13+yrs). The 8-12yrs variant has a minimum score of 0 and a maximum score of 80. The 13+yrs variant has a minimum score of 0 and a maximum score of 88. Mean anxiety scores will be compared across allergic groups.
Food-allergy specific anxiety levels of parents by their child's allergic status, using the Worry About Food Allergy scale | Throughout study, on average 2.5 years
  To determine whether food allergy is associated with changes to food allergy-specific anxiety in the legal caregiver. Food allergy-specific anxiety levels in parents will be assessed using the Worry About Food Allergy Parent scale, which has two variants based on age: one for parents of children aged 8-12yrs and one for parents of children aged 13+yrs. The 8-12yrs variant has a minimum score of 0 and a maximum score of 96. The 13+yrs variant has a minimum score of 0 and a maximum score of 108. Mean anxiety scores will be compared across allergic groups.
Cognitive performance by allergic status, using the Mnemonic Similarity Task | Throughout study, on average 2.5 years
  To determine whether food allergy is associated with changes to cognition in children. Cognition will be measured using the Mnemonic Similarity Task, which assesses a specific form of memory called pattern separation. In this task, participants are assessed on their ability to distinguish 'lure' images (images that are similar but different to images seen in the initial phase) from 'old' images (images that are exactly the same as seen in the initial phase). This ability is recorded as the "Lure Discrimination Index", given on a scale of 0-1, with a higher score indicating great cognitive performance.
General anxiety levels by hippocampal neurogenic dynamics | Throughout study, on average 2.5 years
  To determine whether any observed food allergy-induced changes to hippocampal neurogenesis are linked to changes in general anxiety, as measured by the correlation between mean percentage expression of neurogenic readouts (outlined in Outcomes 1-7) and general anxiety scores (outlined in Outcome 2)
Food allergy-specific anxiety by hippocampal neurogenic dynamics | Throughout study, on average 2.5 years
  To determine whether any observed food allergy-induced changes to hippocampal neurogenesis are linked to changes in food allergy-specific anxiety, as measured by the correlation between mean percentage expression of neurogenic readouts (outlined in Outcomes 1-7) and food allergy-specific anxiety scores (outlined in Outcome 4).
Cognitive performance by hippocampal neurogenic dynamics | Throughout study, on average 2.5 years
  To determine whether any observed food allergy-induced changes to hippocampal neurogenesis are linked to changes in cognitive function, as measured by the correlation between mean percentage expression of neurogenic readouts (outlined in Outcomes 1-7) and cognition scores (outline in Outcome 6)
The association between food allergy diagnosis and Mast Cell Activation (MAT) | Throughout study, on average 2.5 years
  To assess the association between food allergy diagnosis and MAT to specific allergen in this cohort, as measured by mean %CD63 activation of LAD2 mast cells between allergic groups. A higher percentage of %CD63 activation of LAD2 cells indicate a higher allergic response
The association between the Mast Cell Activation (MAT) and hippocampal neurogenesis | Throughout study, on average 2.5 years
  Correlation between %CD63 activation with neurogenesis (Outcomes 1-7)
The association between hippocampal neurogenesis and general anxiety levels | Throughout study, on average 2.5 years
  Correlation between neurogenesis rates (outcomes 1-7) and general anxiety scores (outcome 2)
The association between hippocampal neurogenesis and food allergy-specific anxiety levels | Throughout study, on average 2.5 years
  Correlation between neurogenesis rates (outcomes 1-7) and food allergy-specific anxiety scores (outcome 4)
The association between hippocampal neurogenesis and cognitive performance | Throughout study, on average 2.5 years
  Correlation between neurogenesis rates (outcomes 1-7) and cognitive scores (outcome 6)
The association between hippocampal neurogenesis and food allergy medical history | Throughout study, on average 2.5 years
  To assess the effect of multiple food allergy diagnoses (reported as a number indicated number of other food allergy diagnoses) on hippocampal neurogenesis (outcomes 1-7)
The association between hippocampal neurogenesis and atopic disease diagnoses | Throughout study, on average 2.5 years
  To assess the effect of atopic disease diagnoses (reported as a number indicated number of atopic disease diagnoses) on hippocampal neurogenesis ((outcomes 1-7)

CONTACTS AND LOCATIONS:
Locations (1):
- St Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD